CLINICAL TRIAL: NCT01348490
Title: An Open-Label Assessment of Safety and Efficacy of Ruxolitinib (INCB018424) in Subjects With Primary Myelofibrosis, Post- Essential Thrombocythemia Myelofibrosis, and Post-Polycythemia Vera Myelofibrosis Who Have Platelet Counts of 50 × 10^9/L to 100 × 10^9/L
Brief Title: Ruxolitinib (INCB018424) in Participants With Primary Myelofibrosis (PMF), Post Essential Thrombocythemia-myelofibrosis and Post Polycythemia Vera-myelofibrosis (PPV-MF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB18424-258
Expanded Access: NCT03147742 (Approved for marketing)
Record Dates: First submitted 2011-05-04; First posted 2011-05-05 (Estimated); Results first posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: MPN (Myeloproliferative Neoplasms)
Keywords: PMF; PPV-MF; PET-MF
MeSH Terms: conditions — Myeloproliferative Disorders | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib 5 mg (Experimental): Participants began administration with 5 mg ruxolitinib twice daily (BID) orally. Beginning at the Week 4 visit, doses of ruxolitinib could be increased in 5 mg once a day (QD) increments every 4 weeks every 4 weeks not to exceed a dose of 25 mg BID.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib (INCB018424), 5 mg bid
  Other Names: INCB018424

SUMMARY:
To evaluate the effects of treatment with ruxolitinib (INCB018424) on spleen volume, symptoms and potential side effects in participants with PMF, PPV-MF and PET-MF who have platelet counts of 50 x 10^9/L to 100 x 10^9/L. It is anticipated that individualized dose optimization from the starting ruxolitinib level of 5 mg bid will be associated with reductions in splenomegaly, MF-associated symptoms and inflammatory cytokine levels.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with PMF, PPV-MF or PET-MF as confirmed by bone marrow biopsy
* Discontinuation of all drugs used to treat underlying MF disease at least 14 days prior to baseline visit
* INR <= 1.5 or PTT value < 1.5 x upper limit of normal (ULN) at study entry
* Hemoglobin level at least 6.5 g/dL at Screening visit
* Willingness to be transfused to treat low hemoglobin levels

Exclusion Criteria:

* Females who are pregnant, unable to comply with birth control use to avoid becoming pregnant or breastfeeding
* Males who cannot comply with birth control use to avoid fathering a child
* Platelet count < 50 x10^9/L or absolute neutrophil count (ANC) < 1 x10^9/L at the Screening visit
* Inadequate liver or renal function; Intracranial bleeds or invasive malignancy over the previous 2 years - international normalized ratio (INR) laboratory values cannot be > 1.5 x upper limit of normal at study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2011-06-15 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Langmuir, MD, Study Director — Incyte Corporation
Locations (38):
- United States (38):
  - Birmingham, Alabama
  - Beverly Hills, California
  - Burbank, California
  - La Jolla, California
  - Los Angeles, California
  - Pomona, California
  - San Diego, California
  - New Haven, Connecticut
  - Fort Myers, Florida
  - Jacksonville, Florida
  - Orange City, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Chicago, Illinois
  - Iowa City, Iowa
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Ann Arbor, Michigan
  - Southfield, Michigan
  - St Louis, Missouri
  - Hackensack, New Jersey
  - Morristown, New Jersey
  - Somerville, New Jersey
  - New York, New York
  - Durham, North Carolina
  - Hickory, North Carolina
  - Canton, Ohio
  - Cleveland, Ohio
  - Portland, Oregon
  - Danville, Pennsylvania
  - Hershey, Pennsylvania
  - Charleston, South Carolina
  - Nashville, Tennessee
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Burlington, Vermont

REFERENCES:
- [Derived] Talpaz M, Prchal J, Afrin L, Arcasoy M, Hamburg S, Clark J, Kornacki D, Colucci P, Verstovsek S. Safety and Efficacy of Ruxolitinib in Patients with Myelofibrosis and Low Platelet Counts (50 - 100 x 109/L): Final Analysis of an Open-Label Phase 2 Study. Clin Lymphoma Myeloma Leuk. 2022 May;22(5):336-346. doi: 10.1016/j.clml.2021.10.016. Epub 2021 Nov 2. PMID 34911667
- [Derived] Talpaz M, Paquette R, Afrin L, Hamburg SI, Prchal JT, Jamieson K, Terebelo HR, Ortega GL, Lyons RM, Tiu RV, Winton EF, Natrajan K, Odenike O, Claxton D, Peng W, O'Neill P, Erickson-Viitanen S, Leopold L, Sandor V, Levy RS, Kantarjian HM, Verstovsek S. Interim analysis of safety and efficacy of ruxolitinib in patients with myelofibrosis and low platelet counts. J Hematol Oncol. 2013 Oct 29;6(1):81. doi: 10.1186/1756-8722-6-81. PMID 24283202

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 27 investigative sites in the United States from 15 June 2011 to 19 December 2018.
Pre-assignment Details: A total of 66 participants were enrolled in the study. Fifty-five participants completed 24 weeks of treatment (core treatment period), and 23 participants entered the extension phase.
Groups:
- Ruxolitinib 5 Milligram (mg): Doses may not exceed 10 mg bid except in subjects who continue to meet the above dose escalation criteria, and who have, in addition, a PGIC score of minimally worse, much worse or very much worse while receiving 10 mg bid. Such subjects may continue dose escalation to a maximum dose of 15 mg bid.
  During the extended treatment phase, doses of ruxolitinib may be increased in 5 mg qd increments up to a dose of 25 mg bid if the subject meets the above dose escalation criteria, or per the investigator's discretion.
Period: Overall Study
Arm/Group | Ruxolitinib 5 Milligram (mg)
Started | 66
Completed | 42
Not Completed | 24
Not completed — Death | 1
Not completed — Adverse Event | 3
Not completed — Consent withdrawn | 7
Not completed — Disease progression | 3
Not completed — Lost to Follow-up | 1
Not completed — Termination of clinical trial by sponsor | 1
Not completed — Other Unspecified | 8

BASELINE CHARACTERISTICS:
Population: Safety evaluable population included participants who received at least 1 dose of study drug.
Groups:
- Ruxolitinib 5 mg: Doses may not exceed 10 mg bid except in subjects who continue to meet the above dose escalation criteria, and who have, in addition, a PGIC score of minimally worse, much worse or very much worse while receiving 10 mg bid. Such subjects may continue dose escalation to a maximum dose of 15 mg bid.
  During the extended treatment phase, doses of ruxolitinib may be increased in 5 mg qd increments up to a dose of 25 mg bid if the subject meets the above dose escalation criteria, or per the investigator's discretion.
Arm/Group | Ruxolitinib 5 mg
Number analyzed (Participants) | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.7 (9.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 3
  Ethnicity: Non-Hispanic or Non-Latino | 63
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 58
  Race: Black or African American | 4
  Race: Asian | 2
  Race: Native Hawaiian or Pacific Islander | 1
  Race: Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Spleen Volume at Week 24 by Final Titrated Dose
Description: Magnetic resonance imaging (MRI) of the upper and lower abdomen and pelvis was performed to assess spleen volumes. Computed tomography (CT) scan was performed if participant was not a candidate for MRI or if MRI was not readily available. MRI was performed with a body coil. Spleen volume was obtained by outlining the circumference of the organ and determining the volume using the validated technique of least squares. The MRI (or CT scan in applicable participants) was performed on the first or second day of the baseline period (ie, Day -7 or Day -6), and the site radiologist sent the scan to the central imaging laboratory that same day. The CT scans were processed by the same central laboratory used for MRIs.
Time Frame: Baseline and Week 24
Population: Intent-to-treat (ITT) population included all participants enrolled and treated in the study.
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Groups:
- 5 mg QD or 5 mg BID: Participants received the final titrated dose of ruxolitinib 5 mg QD or 5 mg BID.
- 5 mg AM/ 10 mg PM: Participants received the final titrated dose of ruxolitinib 5 mg AM plus 10 mg PM.
- 10 mg BID: Participants received the final titrated dose of ruxolitinib 10 mg BID.
- 10 mg AM/ 15 mg PM or 15 mg BID: Participants received the final titrated dose of ruxolitinib 10 mg AM plus 15 mg PM or 15 mg BID.
Arm/Group | 5 mg QD or 5 mg BID | 5 mg AM/ 10 mg PM | 10 mg BID | 10 mg AM/ 15 mg PM or 15 mg BID
Number analyzed (Participants) | 16 | 2 | 27 | 6
Percentage change from baseline | -11.6 (18.68) | -17.4 (0.63) | -22.4 (22.86) | -13.4 (22.29)
Statistical Analysis 1: Comparison: 5 mg QD or 5 mg BID; Test type: Other — 1-sample t-test with null hypothesis mean >= 0; p = 0.0250, t-test, 1 sided — 1-sample t-test was used
Statistical Analysis 2: Comparison: 5 mg AM/ 10 mg PM; Test type: Other — 1-sample t-test with null hypothesis mean >= 0; p = 0.0163, t-test, 1 sided — 1-sample t-test was used
Statistical Analysis 3: Comparison: 10 mg BID; Test type: Other — 1-sample t-test with null hypothesis mean >= 0; p < 0.0001, t-test, 1 sided — 1-sample t-test was used
Statistical Analysis 4: Comparison: 10 mg AM/ 15 mg PM or 15 mg BID; Test type: Other — 1-sample t-test with null hypothesis mean >= 0; p = 0.2019, t-test, 1 sided — 1-sample t-test was used

2. Primary Outcome: Percent Change From Baseline in Total Symptom Score (TSS) as Measured by the Modified Myelofibrosis Symptom Assessment Form (MFSAF) V2.0 Diary at Week 24 by Final Titrated Dose
Description: Symptoms of myelofibrosis were assessed using a modified Myelofibrosis Symptom Assessment Form (MFSAF) Version 2.0 diary. Using the diary, patients rated the following symptoms on a scale from 0 (absent) to 10 (worst imaginable): night sweats, itching, abdominal discomfort, pain under ribs on left, feeling of fullness (early satiety), and muscle/bone pain. The total symptom score ranged from 0-60 and was calculated as the sum of the 6 symptom scores. A higher score indicates worse symptoms.
Time Frame: Baseline and Week 24
Population: ITT population included all participants enrolled and treated in the study. For the 5 mg AM/ 10 mg PM arm, the t-test was not calculated due to only having a single participant.
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Arm/Group | 5 mg QD or 5 mg BID | 5 mg AM/ 10 mg PM | 10 mg BID | 10 mg AM/ 15 mg PM or 15 mg BID
Number analyzed (Participants) | 17 | 1 | 29 | 6
Percentage change from baseline | -6.35 (64.207) | -39.51 (NA) — Standard deviation was not calculated due to only having a single participant. | -47.54 (46.886) | 7.95 (113.17)
Statistical Analysis 1: Comparison: 5 mg QD or 5 mg BID; Test type: Other; p = 0.6887, t-test, 1 sided — 1-sample t-test was used
Statistical Analysis 2: Comparison: 10 mg BID; Test type: Other; p < 0.0001, t-test, 1 sided — 1-sample t-test was used
Statistical Analysis 3: Comparison: 10 mg AM/ 15 mg PM or 15 mg BID; Test type: Other; p = 0.8701, t-test, 1 sided — 1-sample t-test was used

3. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAE)
Description: TEAE was defined as adverse events that began or worsened from baseline after the first administration of the study drug.
  Participants were analyzed based on the number of subjects who received a dose within the dose group. The percentages for each column are calculated using this N. Participants who had more than 1 event in an AE category (eg, treatment-related TEAE) are counted once at each dose level the event occurred.
Time Frame: Up to Week 156
Population: Safety evaluable population included participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- >0 - 5 mg: Participants received ruxolitinib up to 0-5mg.
- >5 - 10 mg: Participants received ruxolitinib in the range of 6 mg to 10 mg.
- >10 - 15 mg: Participants received ruxolitinib in the range of 11 to 15 mg.
- >15 - 20 mg: Participants received ruxolitinib in the range of 16 to 20 mg.
- >20 mg: Participants received ruxolitinib, more than 20 mg.
Arm/Group | >0 - 5 mg | >5 - 10 mg | >10 - 15 mg | >15 - 20 mg | >20 mg
Number analyzed (Participants) | 15 | 66 | 54 | 44 | 9
percentage of participants | 93.3 | 74.2 | 61.1 | 77.3 | 55.6

4. Primary Outcome: Percentage of Participants With New Onset Grade 4 Thrombocytopenia Events as Assessed by Common Terminology Criteria for Adverse Events Version 4.03 (CTCAE V4.03)
Description: Participants with platelet count between 50 and 100 × 10^9/L at the screening and/or baseline visit were enrolled in the study. Thrombocytopenia is defined as a condition with low blood platelet count. Grade 4 thrombocytopenia was platelet count < 25 × 10^9/L.
  Participants were analyzed based on the number of subjects who received a dose within the dose group. The percentages for each column are calculated using this N. Participants who had more than 1 event in an AE category (eg, treatment-related TEAE) are counted once at each dose level the event occurred.
Time Frame: Up to Week 156
Population: Safety evaluable population included participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- >0 - 5 mg: Participants received ruxolitinib up to 5 mg.
- >5 - 10 mg: Participants received ruxolitinib in the range of 5 to 10 mg.
- >10 - 15 mg: Participants received ruxolitinib in the range of 10 to 15 mg.
- >15 - 20 mg: Participants received ruxolitinib in the range of 15 to 20 mg.
Arm/Group | >0 - 5 mg | >5 - 10 mg | >10 - 15 mg | >15 - 20 mg | >20 mg
Number analyzed (Participants) | 13 | 66 | 53 | 43 | 8
percentage of participants | 23.1 | 3.0 | 5.7 | 4.7 | 0.0

5. Primary Outcome: Percentage of Participants With New Onset Grade 2 or Higher Hemorrhage as Assessed by CTCAE V4.03
Description: Hemorrhages were defined as any lower level terms by MedDRA included in the Standardized MedDRA Query (SMQ) for hemorrhage terms.
  Participants were analyzed based on the number of subjects who received a dose within the dose group. The percentages for each column are calculated using this N. Participants who had more than 1 event in an AE category (eg, treatment-related TEAE) are counted once at each dose level the event occurred.
Time Frame: Up to Week 156
Population: Safety evaluable population included participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | >0 - 5 mg | >5 - 10 mg | >10 - 15 mg | >15 - 20 mg | >20 mg
Number analyzed (Participants) | 15 | 66 | 54 | 44 | 9
percentage of participants | 6.7 | 3.0 | 1.9 | 2.3 | 11.1

6. Secondary Outcome: Percent Change in Spleen Volume at Week 24 Compared to Baseline
Description: MRI of the upper and lower abdomen and pelvis was performed, to assess spleen volumes. CT scan was performed if participant was not a candidate for MRI, or if MRI was not readily available. MRI was performed with a body coil. Spleen volume was obtained by outlining the circumference of the organ and determining the volume using the validated technique of least squares. The MRI (or CT scan in applicable participants) was performed on the first or second day of the baseline period (ie, Day -7 or Day -6), and the site radiologist sent the scan to the central imaging laboratory that same day. The CT scans were processed by the same central laboratory used for MRIs.
Time Frame: Baseline and Week 24
Population: ITT population included all participants enrolled and treated in the study.
Measure: Mean (Standard Deviation); unit: Percentage
Groups:
- Ruxolitinib: Participants who received ruxolitinib doses as 5 mg QD or 5 mg BID, 5 mg AM/ 10 mg PM, 10 mg BID, and 10 mg AM/ 15 mg PM or 15 mg BID.
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 51
Percentage | -17.8 (21.27)
Statistical Analysis 1: Comparison: Ruxolitinib; Test type: Other; p < 0.0001, t-test, 1 sided — 1-sample t-test was used

7. Secondary Outcome: Percent Change in Total Symptom Score as Measured by the Modified MFSAF V2.0 Diary at Week 24 Compared to Baseline
Description: as for outcome 2
Time Frame: Baseline and Week 24
Population: ITT population included all participants enrolled and treated in the study.
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 53
Percentage change from baseline | -27.90 (64.818)
Statistical Analysis 1: Comparison: Ruxolitinib; Test type: Other; p = 0.0028, t-test, 1 sided — 1-sample t-test was used

8. Secondary Outcome: Percentage of Participants With ≥ 35% Reduction in Spleen Volume at Week 24 Compared to Baseline
Description: MRI of the upper and lower abdomen and pelvis was performed, to assess spleen volumes. CT scan was performed if participant is not a candidate for MRI, or if MRI is not readily available. MRI was performed with a body coil. Spleen volume was obtained by outlining the circumference of the organ and determining the volume using the validated technique of least squares. The MRI (or CT scan in applicable participants) was performed on the first or second day of the baseline period (ie, Day -7 or Day -6), and the site radiologist sent the scan to the central imaging laboratory that same day. The CT scans were processed by the same central laboratory used for MRIs.
Time Frame: Baseline and Week 24
Population: Efficacy evaluable participants included all participants enrolled and treated in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 5 mg QD or 5 mg BID | 5 mg AM/ 10 mg PM | 10 mg BID | 10 mg AM/ 15 mg PM or 15 mg BID
Number analyzed (Participants) | 21 | 3 | 33 | 7
percentage of participants | 4.8 [0.1 to 23.8] | 0.0 [0.0 to 70.8] | 24.2 [11.1 to 42.3] | 28.6 [3.7 to 71.0]

9. Secondary Outcome: Percentage of Participants With ≥10% Reduction in Spleen Volume at Week 24 Compared to Baseline
Description: as for outcome 8
Time Frame: Baseline and Week 24
Population: Efficacy evaluable participants included all participants enrolled and treated in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 5 mg QD or 5 mg BID | 5 mg AM/ 10 mg PM | 10 mg BID | 10 mg AM/ 15 mg PM or 15 mg BID
Number analyzed (Participants) | 21 | 3 | 33 | 7
percentage of participants | 42.9 [21.8 to 66.0] | 66.7 [9.4 to 99.2] | 63.6 [45.1 to 79.6] | 28.6 [3.7 to 71.0]

10. Secondary Outcome: Percentage of Participants With ≥ 50% Improvement in Total Symptom Score as Measured by the Modified MFSAF V2.0 Diary at Week 24 Compared to Baseline
Description: as for outcome 2
Time Frame: Baseline and Week 24
Population: Efficacy evaluable participants included all participants enrolled and treated in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 5 mg QD or 5 mg BID | 5 mg AM/ 10 mg PM | 10 mg BID | 10 mg AM/ 15 mg PM or 15 mg BID
Number analyzed (Participants) | 21 | 3 | 34 | 7
percentage of participants | 28.6 [11.3 to 52.2] | 0.0 [0.0 to 70.8] | 44.1 [27.2 to 62.1] | 28.6 [3.7 to 71.0]

11. Secondary Outcome: Change in Spleen Length Measured by Palpation
Description: Measurement of spleen length below the left costal margin was measured by palpation at each study visit. Investigators were provided with a soft centimeter ruler so that palpable spleen length was measured in centimeters and not in finger breadths. The edge of the spleen was determined by palpation, and measured in centimeters, using a soft ruler, from the costal margin to the point of greatest splenic protrusion.
Time Frame: Up to Week 156
Population: Efficacy evaluable participants included all participants enrolled and treated in the study. 'Number Analyzed' is number of participants with data available at a particular time point.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | 5 mg QD or 5 mg BID | 5 mg AM/ 10 mg PM | 10 mg BID | 10 mg AM/ 15 mg PM or 15 mg BID
Number analyzed (Participants) | 21 | 4 | 34 | 7
cm
  Baseline: number analyzed (Participants) | 21 | 3 | 32 | 7
  Baseline | 11.48 (5.810) | 14.00 (4.359) | 13.13 (8.241) | 14.71 (6.726)
  Change at Week 4: number analyzed (Participants) | 20 | 3 | 31 | 6
  Change at Week 4 | -3.40 (3.068) | -4.00 (6.083) | -1.84 (3.195) | 0.00 (3.688)
  Change at Week 8: number analyzed (Participants) | 20 | 3 | 32 | 7
  Change at Week 8 | -4.65 (3.558) | -5.33 (4.933) | -2.81 (3.514) | -1.14 (2.340)
  Change at Week 12: number analyzed (Participants) | 19 | 2 | 31 | 7
  Change at Week 12 | -4.53 (4.812) | -6.50 (3.536) | -3.74 (5.118) | -3.71 (7.544)
  Change at Week 16: number analyzed (Participants) | 19 | 2 | 29 | 7
  Change at Week 16 | -3.79 (4.973) | -4.50 (3.536) | -3.69 (4.343) | -2.00 (2.449)
  Change at Week 20: number analyzed (Participants) | 16 | 2 | 29 | 6
  Change at Week 20 | -4.56 (4.844) | -7.50 (4.950) | -5.28 (5.567) | -3.50 (7.064)
  Change at Week 24: number analyzed (Participants) | 16 | 2 | 28 | 6
  Change at Week 24 | -4.25 (5.092) | -7.00 (5.657) | -4.57 (5.541) | -1.33 (3.983)
  Change at Week 36: number analyzed (Participants) | 1 | 1 | 4 | 1
  Change at Week 36 | -7.00 (NA) — Standard deviation was not estimated due to less number of participants. | -11.00 (NA) — Standard deviation was not estimated due to less number of participants. | -2.75 (3.862) | 1.00 (NA) — Standard deviation was not estimated due to less number of participants.
  Change at Week 48: number analyzed (Participants) | 1 | 1 | 3 | 2
  Change at Week 48 | -7.00 (NA) — Standard deviation was not estimated due to less number of participants. | -11.00 (NA) — Standard deviation was not estimated due to less number of participants. | -2.33 (2.517) | 0.00 (0.000)
  Change at Week 60: number analyzed (Participants) | 1 | 1 | 3 | 2
  Change at Week 60 | -7.00 (NA) — Standard deviation was not estimated due to less number of participants. | -11.00 (NA) — Standard deviation was not estimated due to less number of participants. | -2.67 (2.517) | 1.50 (2.121)
  Change at Week 72: number analyzed (Participants) | 1 | 1 | 2 | 1
  Change at Week 72 | -4.00 (NA) — Standard deviation was not estimated due to less number of participants. | -11.00 (NA) — Standard deviation was not estimated due to less number of participants. | -1.50 (2.121) | 1.00 (NA) — Standard deviation was not estimated due to less number of participants.
  Change at Week 84: number analyzed (Participants) | 1 | 0 | 1 | 1
  Change at Week 84 | -4.00 (NA) — Standard deviation was not estimated due to less number of participants. |  | -3.00 (NA) — Standard deviation was not estimated due to less number of participants. | -2.00 (NA) — Standard deviation was not estimated due to less number of participants.
  Change at Week 96: number analyzed (Participants) | 1 | 1 | 1 | 0
  Change at Week 96 | -4.00 (NA) — Standard deviation was not estimated due to less number of participants. | -8.00 (NA) — Standard deviation was not estimated due to less number of participants. | 0.00 (NA) — Standard deviation was not estimated due to less number of participants. |
  Change at Week 108: number analyzed (Participants) | 1 | 1 | 1 | 0
  Change at Week 108 | -4.00 (NA) — Standard deviation was not estimated due to less number of participants. | -10.00 (NA) — Standard deviation was not estimated due to less number of participants. | 0.00 (NA) — Standard deviation was not estimated due to less number of participants. |
  Change at Week 120: number analyzed (Participants) | 1 | 1 | 1 | 0
  Change at Week 120 | -4.00 (NA) — Standard deviation was not estimated due to less number of participants. | -6.00 (NA) — Standard deviation was not estimated due to less number of participants. | 2.00 (NA) — Standard deviation was not estimated due to less number of participants. |
  Change at Week 132: number analyzed (Participants) | 1 | 1 | 1 | 0
  Change at Week 132 | -4.00 (NA) — Standard deviation was not estimated due to less number of participants. | -5.00 (NA) — Standard deviation was not estimated due to less number of participants. | 1.00 (NA) — Standard deviation was not estimated due to less number of participants. |
  Change at Week 144: number analyzed (Participants) | 1 | 1 | 1 | 0
  Change at Week 144 | -4.00 (NA) — Standard deviation was not estimated due to less number of participants. | -3.00 (NA) — Standard deviation was not estimated due to less number of participants. | 0.00 (NA) — Standard deviation was not estimated due to less number of participants. |
  Change at Week 156: number analyzed (Participants) | 1 | 1 | 1 | 0
  Change at Week 156 | -4.00 (NA) — Standard deviation was not estimated due to less number of participants. | -3.00 (NA) — Standard deviation was not estimated due to less number of participants. | 0.00 (NA) — Standard deviation was not estimated due to less number of participants. |

12. Secondary Outcome: Percent Change From Baseline in Spleen Length Measured by Palpation
Description: as for outcome 11
Time Frame: Up to Week 156
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | 5 mg QD or 5 mg BID | 5 mg AM/ 10 mg PM | 10 mg BID | 10 mg AM/ 15 mg PM or 15 mg BID
Number analyzed (Participants) | 21 | 4 | 34 | 7
Percentage
  Percent Change at Week 4: number analyzed (Participants) | 19 | 3 | 28 | 5
  Percent Change at Week 4 | -38.61 (36.532) | -26.62 (36.906) | -21.88 (33.800) | -1.42 (22.902)
  Percent Change at Week 8: number analyzed (Participants) | 19 | 3 | 29 | 6
  Percent Change at Week 8 | -50.64 (39.930) | -37.95 (28.772) | -28.32 (31.151) | -8.72 (13.991)
  Percent Change at Week 12: number analyzed (Participants) | 18 | 2 | 28 | 6
  Percent Change at Week 12 | -49.90 (48.623) | -50.35 (8.348) | -38.21 (39.936) | -22.41 (40.833)
  Percent Change at Week 16: number analyzed (Participants) | 18 | 2 | 26 | 6
  Percent Change at Week 16 | -43.24 (48.173) | -32.99 (15.222) | -38.67 (36.070) | -14.33 (14.903)
  Percent Change at Week 20: number analyzed (Participants) | 15 | 2 | 26 | 5
  Percent Change at Week 20 | -44.58 (46.490) | -56.60 (17.187) | -48.06 (38.826) | -27.75 (39.024)
  Percent Change at Week 24: number analyzed (Participants) | 15 | 2 | 25 | 5
  Percent Change at Week 24 | -45.39 (53.913) | -51.04 (25.043) | -42.01 (36.899) | -9.89 (25.001)
  Percent Change at Week 36: number analyzed (Participants) | 1 | 1 | 3 | 1
  Percent Change at Week 36 | -58.33 (NA) — Standard deviation was not estimated due to less number of participants. | -68.75 (NA) — Standard deviation was not estimated due to less number of participants. | -20.76 (27.637) | 5.00 (NA) — Standard deviation was not estimated due to less number of participants.
  Percent Change at Week 48: number analyzed (Participants) | 1 | 1 | 2 | 1
  Percent Change at Week 48 | -58.33 (NA) — Standard deviation was not estimated due to less number of participants. | -68.75 (NA) — Standard deviation was not estimated due to less number of participants. | -31.82 (19.285) | 0.00 (NA) — Standard deviation was not estimated due to less number of participants.
  Percent Change at Week 60: number analyzed (Participants) | 1 | 1 | 2 | 1
  Percent Change at Week 60 | -58.33 (NA) — Standard deviation was not estimated due to less number of participants. | -68.75 (NA) — Standard deviation was not estimated due to less number of participants. | -36.36 (12.856) | 15.00 (NA) — Standard deviation was not estimated due to less number of participants.
  Percent Change at Week 72: number analyzed (Participants) | 1 | 1 | 1 | 1
  Percent Change at Week 72 | -33.33 (NA) — Standard deviation was not estimated due to less number of participants. | -68.75 (NA) — Standard deviation was not estimated due to less number of participants. | -27.27 (NA) — Standard deviation was not estimated due to less number of participants. | 5.00 (NA) — Standard deviation was not estimated due to less number of participants.
  Percent Change at Week 84: number analyzed (Participants) | 1 | 0 | 1 | 1
  Percent Change at Week 84 | -33.33 (NA) — Standard deviation was not estimated due to less number of participants. |  | -27.27 (NA) — Standard deviation was not estimated due to less number of participants. | -10.00 (NA) — Standard deviation was not estimated due to less number of participants.
  Percent Change at Week 96: number analyzed (Participants) | 1 | 1 | 0 | 0
  Percent Change at Week 96 | -33.33 (NA) — Standard deviation was not estimated due to less number of participants. | -50.00 (NA) — Standard deviation was not estimated due to less number of participants. |  |
  Percent Change at Week 108: number analyzed (Participants) | 1 | 1 | 0 | 0
  Percent Change at Week 108 | -33.33 (NA) — Standard deviation was not estimated due to less number of participants. | -62.50 (NA) — Standard deviation was not estimated due to less number of participants. |  |
  Percent Change at Week 120: number analyzed (Participants) | 1 | 1 | 0 | 0
  Percent Change at Week 120 | -33.33 (NA) — Standard deviation was not estimated due to less number of participants. | -37.50 (NA) — Standard deviation was not estimated due to less number of participants. |  |
  Percent Change at Week 132: number analyzed (Participants) | 1 | 1 | 0 | 0
  Percent Change at Week 132 | -33.33 (NA) — Standard deviation was not estimated due to less number of participants. | -31.25 (NA) — Standard deviation was not estimated due to less number of participants. |  |
  Percent Change at Week 144: number analyzed (Participants) | 1 | 1 | 0 | 0
  Percent Change at Week 144 | -33.33 (NA) — Standard deviation was not estimated due to less number of participants. | -18.75 (NA) — Standard deviation was not estimated due to less number of participants. |  |
  Percent Change at Week 156: number analyzed (Participants) | 1 | 1 | 0 | 0
  Percent Change at Week 156 | -33.33 (NA) — Standard deviation was not estimated due to less number of participants. | -18.75 (NA) — Standard deviation was not estimated due to less number of participants. |  |

13. Secondary Outcome: Patient Global Impression of Change (PGIC) Score at Each Visit
Description: Symptoms of myelofibrosis were assessed using the PGIC questionnaire. Using the questionnaire, patients rated the overall sense of treatment effect on their symptoms on a scale of 1 (very much improved)- 7(very much worse). The specific wording was: Since the start of the treatment you've received in this study, your myelofibrosis symptoms are: 1) Very much improved, 2) Much improved, 3) Minimally improved, 4) No change, 5) Minimally worse, 6) Much worse, 7) Very much worse. A higher score indicates worse symptoms.
Time Frame: Up to Week 156
Population: Efficacy evaluable participants included all participants enrolled and treated in the study. 'Number Analyzed' is number of participants with data available at the particular time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 5 mg QD or 5 mg BID | 5 mg AM/ 10 mg PM | 10 mg BID | 10 mg AM/ 15 mg PM or 15 mg BID
Number analyzed (Participants) | 21 | 4 | 34 | 7
score on a scale
  Week 4: number analyzed (Participants) | 20 | 4 | 33 | 7
  Week 4 | 2.8 (0.89) | 2.8 (1.26) | 2.6 (1.09) | 3.3 (0.76)
  Week 8: number analyzed (Participants) | 20 | 4 | 33 | 7
  Week 8 | 2.7 (1.22) | 2.3 (0.96) | 2.2 (0.99) | 2.9 (0.69)
  Week 12: number analyzed (Participants) | 19 | 3 | 33 | 7
  Week 12 | 2.4 (0.96) | 2.3 (1.15) | 2.2 (1.17) | 3.4 (1.27)
  Week 16: number analyzed (Participants) | 19 | 3 | 30 | 7
  Week 16 | 2.4 (0.83) | 2.0 (1.00) | 1.9 (0.91) | 3.3 (0.95)
  Week 20: number analyzed (Participants) | 17 | 3 | 29 | 6
  Week 20 | 2.4 (0.86) | 2.3 (0.58) | 1.9 (1.11) | 2.3 (0.82)
  Week 24: number analyzed (Participants) | 17 | 3 | 30 | 5
  Week 24 | 2.9 (1.27) | 2.3 (0.58) | 1.9 (0.98) | 2.0 (1.00)
  Week 36: number analyzed (Participants) | 1 | 1 | 4 | 2
  Week 36 | 2.0 (NA) — Standard deviation was not estimated due to less number of participants. | 3.0 (NA) — Standard deviation was not estimated due to less number of participants. | 1.8 (0.50) | 2.5 (0.71)
  Week 48: number analyzed (Participants) | 0 | 2 | 3 | 2
  Week 48 |  | 2.5 (0.71) | 1.3 (0.58) | 2.0 (0.00)
  Week 60: number analyzed (Participants) | 1 | 2 | 3 | 2
  Week 60 | 2.0 (NA) — Standard deviation was not estimated due to less number of participants. | 2.5 (0.71) | 1.7 (0.58) | 3.0 (0.00)
  Week 72: number analyzed (Participants) | 1 | 2 | 0 | 1
  Week 72 | 2.0 (NA) — Standard deviation was not estimated due to less number of participants. | 2.5 (0.71) |  | 4.0 (NA) — Standard deviation was not estimated due to less number of participants.
  Week 84: number analyzed (Participants) | 0 | 1 | 2 | 1
  Week 84 |  | 2.0 (NA) — Standard deviation was not estimated due to less number of participants. | 1.0 (0.00) | 3.0 (NA) — Standard deviation was not estimated due to less number of participants.
  Week 96: number analyzed (Participants) | 1 | 2 | 0 | 0
  Week 96 | 2.0 (NA) — Standard deviation was not estimated due to less number of participants. | 2.5 (0.71) |  |
  Week 108: number analyzed (Participants) | 1 | 2 | 1 | 0
  Week 108 | 2.0 (NA) — Standard deviation was not estimated due to less number of participants. | 2.5 (0.71) | 1.0 (NA) — Standard deviation was not estimated due to less number of participants. |
  Week 120: number analyzed (Participants) | 1 | 2 | 0 | 0
  Week 120 | 2.0 (NA) — Standard deviation was not estimated due to less number of participants. | 2.5 (0.71) |  |
  Week 132: number analyzed (Participants) | 1 | 2 | 1 | 0
  Week 132 | 2.0 (NA) — Standard deviation was not estimated due to less number of participants. | 3.0 (1.41) | 1.0 (NA) — Standard deviation was not estimated due to less number of participants. |
  Week 144: number analyzed (Participants) | 1 | 2 | 1 | 0
  Week 144 | 2.0 (NA) — Standard deviation was not estimated due to less number of participants. | 2.5 (0.71) | 1.0 (NA) — Standard deviation was not estimated due to less number of participants. |
  Week 156: number analyzed (Participants) | 1 | 2 | 1 | 0
  Week 156 | 2.0 (NA) — Standard deviation was not estimated due to less number of participants. | 3.0 (1.41) | 1.0 (NA) — Standard deviation was not estimated due to less number of participants. |

ADVERSE EVENTS:
Time Frame: Up to approximately 161 weeks
Description: Safety evaluable population included participants who received at least 1 dose of study drug. Data for adverse events was reported as per the total daily dose the participant was receiving at the time of the event.
Arm/Group | >0 - 5 mg | >5 - 10 mg | >10 - 15 mg | >15 - 20 mg | >20 mg
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/66 | 0/54 | 2/44 | 0/9
Serious Adverse Events (participants affected / at risk) | 5/15 | 8/66 | 4/54 | 9/44 | 1/9
Other Adverse Events (participants affected / at risk) | 13/15 | 43/66 | 26/54 | 31/44 | 5/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | >0 - 5 mg (N=15) | >5 - 10 mg (N=66) | >10 - 15 mg (N=54) | >15 - 20 mg (N=44) | >20 mg (N=9)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 1 | 0 — General disorders and administration site conditions
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 1 | 1
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Hypnagogic hallucination (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Epididymitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | >0 - 5 mg (N=15) | >5 - 10 mg (N=66) | >10 - 15 mg (N=54) | >15 - 20 mg (N=44) | >20 mg (N=9)
Anaemia (Blood and lymphatic system disorders) | 3 | 7 | 4 | 5 | 0
Reticulocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 11 | 4 | 2 | 1
Cardiomegaly (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
Cyanosis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 4 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 1 | 0 | 0 | 0
Scleral haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 3 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 4 | 2 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 7 | 7 | 3 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 6 | 2 | 4 | 0
Vomiting (Gastrointestinal disorders) | 2 | 3 | 0 | 3 | 0
Asthenia (General disorders) | 0 | 0 | 4 | 0 | 0 — General disorders and administration site conditions
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 1 — General disorders and administration site conditions
Early satiety (General disorders) | 0 | 2 | 0 | 0 | 1 — General disorders and administration site conditions
Fatigue (General disorders) | 2 | 7 | 5 | 3 | 1 — General disorders and administration site conditions
Oedema (General disorders) | 1 | 2 | 1 | 0 | 0 — General disorders and administration site conditions
Oedema peripheral (General disorders) | 1 | 9 | 4 | 6 | 0 — General disorders and administration site conditions
Pain (General disorders) | 1 | 1 | 0 | 0 | 0 — General disorders and administration site conditions
Pyrexia (General disorders) | 1 | 0 | 3 | 3 | 1 — General disorders and administration site conditions
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Gallbladder disorder (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 1 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 2 | 6 | 1
Vaginal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 5 | 3 | 2 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Blast cell count increased (Investigations) | 1 | 1 | 1 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood creatinine decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Cardioactive drug level increased (Investigations) | 1 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 1 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 3 | 0
Occult blood positive (Investigations) | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 3 | 3 | 3 | 0
Serum ferritin increased (Investigations) | 1 | 1 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 1 | 1 | 0 | 1 | 0
White blood cell count increased (Investigations) | 1 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 1 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 2 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 3 | 1 | 3 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Iron overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 1 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 3 | 0 | 3 | 1
Headache (Nervous system disorders) | 0 | 4 | 3 | 2 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Urine flow decreased (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 4 | 0 | 2 | 2
Hypertension (Vascular disorders) | 1 | 2 | 0 | 2 | 1

LIMITATIONS AND CAVEATS:
Participants with platelet counts of 50 to 100 x 10^9/L were enrolled to begin ruxolitinib at 5 mg BID. Subjects could then titrate their dose to an dose that offers benefit. Only the overall data was calculated for the Participant and Baseline data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement

DOCUMENTS (2):
  • Study Protocol (2013-08-09): https://cdn.clinicaltrials.gov/large-docs/90/NCT01348490/Prot_000.pdf
  • Statistical Analysis Plan (2012-01-17): https://cdn.clinicaltrials.gov/large-docs/90/NCT01348490/SAP_001.pdf